CLINICAL TRIAL: NCT04502784
Title: Investigation of the Mechanisms for the Development of Hypophosphataemia Following Administration of Intravenous Iron in Patients With Severe Anaemia
Brief Title: Investigation of Hypophosphataemia Following Intravenous Iron
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Belfast Health and Social Care Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 18195BR-SS
Record Dates: First submitted 2020-08-04; First posted 2020-08-06 (Actual); Last update posted 2020-08-06 (Actual); Status verified 2020-08

CONDITIONS: Hypophosphatemia; Chronic Kidney Diseases; Intestinal Disease; Anemia
MeSH Terms: conditions — Hypophosphatemia; Renal Insufficiency, Chronic; Intestinal Diseases; Anemia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum, EDTA plasma, and urine samples will be collected and stored for batch analysis.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Chronic Kidney Disease: This group will consist of 10 patients who have previously been diagnosed with chronic kidney disease and are receiving intravenous iron due to anaemia.
- Intestinal failure: This group will consist of 10 patients who have previously been diagnosed with intestinal conditions and are receiving intravenous iron due to anaemia.
- Healthy Volunteers: This group will consist of 20 healthy volunteers. This group will act as a comparator for the CKD and intestinal failure groups.

SUMMARY:
Anaemia (low haemoglobin levels) can develop in a number of conditions, including chronic kidney disease (CKD) and intestinal conditions (e.g. inflammatory bowel disease, intestinal failure). Intravenous iron can be given to patients with these conditions to help correct their aneaemia. However, intravenous iron has been associated with the development of low phosphate levels - hypophophosphataemia. The aim of this study is to determine potential causes of hypophosphataemia following administration of intravenous iron.

DETAILED DESCRIPTION:
Low levels of iron can lead to anaemia, known as iron deficiency anaemia, which can be debilitating due to symptoms such as shortness of breath, fatigue, and dizziness. Iron deficiency anaemia can be treated by giving iron supplementation. Iron supplements can be taken orally or can be given intravenously (through the veins). Giving iron intravenously has advantages over iron supplements taken orally, which can cause side effects such as stomach pain and cramping. However, giving iron intravenously has been associated with the development of low levels of phosphate in the blood. This is known as hypophosphataemia. Phosphate is an important salt in the body and has a number of important functions. Very low levels of phosphate can cause muscle pain, disorientation, seizures and heart problems. It is unclear why giving iron intravenously can cause hypophosphataemia. This project aims to investigate the potential causes of hypophosphataemia in patients who receive intravenous iron as treatment for anaemia associated with their condition. Patients with chronic kidney disease (CKD) and intestinal failure will be recruited to the study, since people with CKD may handle iron differently than those with healthy kidneys. Samples will be taken at two time points: prior to giving the intravenous iron and at the patient's next appointment. Healthy volunteers will also be recruited to the study to allow comparison between the groups receiving iron and those who do not receive iron. Samples will be analysed to determine potential causes of hypophosphataemia. Results from before and after iron is given will be compared to determine if any of the participants developed hypophosphataemia and if any other test are affected which may explain why this has developed.

ELIGIBILITY:
Inclusion Criteria:

For Patients

* aged 18 years or older
* previously diagnosed with intestinal failure or advanced CKD
* have anaemia requiring administration of intravenous iron
* be able to adequately speak and understand English
* Have capacity to give written informed consent

For Healthy Volunteers

* aged 18 years or more
* be able to adequately speak and understand English
* have capacity to give written informed consent

Exclusion Criteria:

For patients

* have dialysis-dependent CKD
* participation in any other study which will affect results of the current study

For Healthy Volunteers

* have CKD (eGFR <60 mls/min/1.73^2)
* history of any form of metabolic bone disease
* Participation in any other study which will affect the results of the current study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with intestinal failure or CKD will be recruited from iron infusion clinics, which are based in secondary care. Healthy Volunteers will be recruited from laboratory staff from within the Belfast Health and Social Care Trust
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2019-10-07 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
FGF23 levels before and after intravenous iron | 8 weeks
  Measurement of FGF23 levels in patients with CKD before and after intravenous iron administration

SECONDARY OUTCOMES:
FGF23 levels in patients with CKD and healthy volunteers | 1 week
  Comparison of measured FGF23 levels in patients with CKD and healthy volunteers
Characterisation of pre-analytical factors affecting FGF23 levels | 1 week
  To examine the effect of delayed separation and fasting vs non-fasting on FGF23 levels

CONTACTS AND LOCATIONS:
Overall Officials: Brona Roberts, Principal Investigator — Beflast Health and Social Care Trust
Locations (1):
- Belfast Health and Social Care Trust, Belfast, United Kingdom

IPD SHARING:
Plan to Share IPD: No